CLINICAL TRIAL: NCT01140282
Title: Combined Exercise Program for Early Breast Cancer Survivors
Brief Title: Exercise Program for Early Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1B-12-1; NCI-2010-01265
Record Dates: First submitted 2010-06-04; First posted 2010-06-09 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
Keywords: cancer survivor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Control) (Active Comparator): Patients refrain from increasing physical activity levels for 16 weeks.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment; Procedure: management of therapy complications
- Arm II (Exercise) (Experimental): Patients participate in supervised exercise sessions over 60 minutes thrice weekly and are encouraged to participate in a home-based exercise session over 30-45 minutes once weekly for 16 weeks.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment; Procedure: management of therapy complications; Behavioral: exercise intervention

INTERVENTIONS:
Other: questionnaire administration — Administered within 3 days of baseline testing and at post-trial visit
Procedure: quality-of-life assessment — Administered within 3 days of baseline testing and at post-trial visit
  Other Names: quality of life assessment
Procedure: management of therapy complications — Assessed within 3 days of baseline testing and at post-trial visit
  Other Names: complications of therapy, management of
Behavioral: exercise intervention — 12 week exercise intervention
  Arms: Arm II (Exercise)

SUMMARY:
Rationale: Exercise therapy may improve the quality of life of breast cancer survivors.

Purpose: This randomized clinical trial studies exercise therapy and quality of life in postmenopausal early breast cancer survivors receiving aromatase inhibitor therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether a 16-week exercise intervention will improve components of metastasis (MetS) in breast cancer survivors soon after completion of cancer-related treatments by measuring changes in body composition, waist circumference, blood pressure, and serum levels of insulin, glucose, lipids, C-reactive protein, and hemoglobin A1c (HbA1c).

II. To determine whether a 16-week exercise intervention will improve physical fitness in breast cancer survivors soon after completion of cancer-related treatments by measuring cardiorespiratory fitness and muscle strength.

III. To assesses the feasibility of a supervised exercise intervention in early breast cancer survivors.

IV. To determine whether a 16-week exercise intervention will result in a reduction in adipose tissue inflammation in obese breast cancer survivors soon after completion of cancer-related treatments by measuring ATM phenotype and ATM cytokine expression.

V. To determine whether breast cancer survivors can maintain positive benefits of an exercise intervention following a 12-week follow-up period by measuring changes in body composition, waist circumference, blood pressure, and serum levels of insulin, glucose, lipids, C-reactive protein, and HbA1c, cardiorespiratory fitness and muscle strength.

OUTLINE:

Patients are randomized to 1 of 2 arms.

Arm I (Control): Patients refrain from increasing physical activity levels for 16 weeks.

Arm II (Exercise): Patients participate in supervised exercise sessions over 60 minutes thrice weekly and are encouraged to participate in a home-based exercise session over 30-45 minutes once weekly for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (I-III) with a first primary invasive breast cancer
* Have undergone a lumpectomy or mastectomy
* Have completed neoadjuvant/adjuvant chemotherapy and able to initiate Exercise program (if randomized to that arm) within 12 weeks of therapy completion
* Body mass index (BMI) > 25 kg/m^2 or body fat > 30% (determined by Dr. Dieli-Conwright at baseline visit)
* Currently participate in less than 60 minutes of physical activity per week May use adjuvant endocrine therapy if use will be continued for duration of study period
* Nonsmokers (i.e., not smoking during previous 12 months)
* Willing to travel to the exercise facility and USC
* Able to provide physician clearance to participate in exercise program
* Women of all racial and ethnic backgrounds will be included in the study enrollment process

Exclusion Criteria:

* History of chronic disease including diabetes, uncontrolled hypertension or thyroid disease
* Weight reduction >= 10% within past 6 months
* Diagnosed with human epidermal growth factor receptor 2 (HER2)-positive tumor (exclusion due to patient use of Herceptin medication for 1 year following chemotherapy)
* Metastatic disease
* Planned reconstructive surgery with flap repair during trial and follow-up period
* Cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in body composition, waist circumference, blood pressure, and serum levels of insulin, glucose, lipids, C-reactive protein, and HbA1c | At week 16
Improvement of physical fitness, cardiorespiratory fitness, and muscle strength | At week 16
Feasibility of a supervised exercise program for cancer survivors | At week 16
Maintain positive benefits of an exercise intervention | 12 weeks post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Dieli-Conwright CM, Sami N, Norris MK, Wan J, Kumagai H, Kim SJ, Cohen P. Effect of aerobic and resistance exercise on the mitochondrial peptide MOTS-c in Hispanic and Non-Hispanic White breast cancer survivors. Sci Rep. 2021 Aug 19;11(1):16916. doi: 10.1038/s41598-021-96419-z. PMID 34413391
- [Derived] Dieli-Conwright CM, Courneya KS, Demark-Wahnefried W, Sami N, Norris MK, Fox FS, Buchanan TA, Spicer D, Bernstein L, Tripathy D. Aerobic and resistance exercise improve patient-reported sleep quality and is associated with cardiometabolic biomarkers in Hispanic and non-Hispanic breast cancer survivors who are overweight or obese: results from a secondary analysis. Sleep. 2021 Oct 11;44(10):zsab111. doi: 10.1093/sleep/zsab111. PMID 33929533
- [Derived] Lee K, Sami N, Tripathy D, Demark-Wahnefried W, Norris MK, Courneya KS, Dieli-Conwright CM. Aerobic and resistance exercise improves Reynolds risk score in overweight or obese breast cancer survivors. Cardiooncology. 2020 Nov 24;6(1):27. doi: 10.1186/s40959-020-00084-6. PMID 33292676
- [Derived] Sweeney FC, Demark-Wahnefried W, Courneya KS, Sami N, Lee K, Tripathy D, Yamada K, Buchanan TA, Spicer DV, Bernstein L, Mortimer JE, Dieli-Conwright CM. Aerobic and Resistance Exercise Improves Shoulder Function in Women Who Are Overweight or Obese and Have Breast Cancer: A Randomized Controlled Trial. Phys Ther. 2019 Oct 28;99(10):1334-1345. doi: 10.1093/ptj/pzz096. PMID 31309977
- [Derived] Lee K, Tripathy D, Demark-Wahnefried W, Courneya KS, Sami N, Bernstein L, Spicer D, Buchanan TA, Mortimer JE, Dieli-Conwright CM. Effect of Aerobic and Resistance Exercise Intervention on Cardiovascular Disease Risk in Women With Early-Stage Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2019 May 1;5(5):710-714. doi: 10.1001/jamaoncol.2019.0038. PMID 30920602
- [Derived] Dieli-Conwright CM, Courneya KS, Demark-Wahnefried W, Sami N, Lee K, Sweeney FC, Stewart C, Buchanan TA, Spicer D, Tripathy D, Bernstein L, Mortimer JE. Aerobic and resistance exercise improves physical fitness, bone health, and quality of life in overweight and obese breast cancer survivors: a randomized controlled trial. Breast Cancer Res. 2018 Oct 19;20(1):124. doi: 10.1186/s13058-018-1051-6. PMID 30340503
- [Derived] Dieli-Conwright CM, Courneya KS, Demark-Wahnefried W, Sami N, Lee K, Buchanan TA, Spicer DV, Tripathy D, Bernstein L, Mortimer JE. Effects of Aerobic and Resistance Exercise on Metabolic Syndrome, Sarcopenic Obesity, and Circulating Biomarkers in Overweight or Obese Survivors of Breast Cancer: A Randomized Controlled Trial. J Clin Oncol. 2018 Mar 20;36(9):875-883. doi: 10.1200/JCO.2017.75.7526. Epub 2018 Jan 22. PMID 29356607
- [Derived] Dieli-Conwright CM, Mortimer JE, Schroeder ET, Courneya K, Demark-Wahnefried W, Buchanan TA, Tripathy D, Bernstein L. Randomized controlled trial to evaluate the effects of combined progressive exercise on metabolic syndrome in breast cancer survivors: rationale, design, and methods. BMC Cancer. 2014 Apr 3;14:238. doi: 10.1186/1471-2407-14-238. PMID 24708832